CLINICAL TRIAL: NCT05913284
Title: Intravenous Methadone in Perioperative Acute and Chronic Management in Chinese Adult Cardiac Surgical Patients: a Pilot Randomized Controlled Trial
Brief Title: Intravenous Methadone in Perioperative Acute and Chronic Management in Chinese Adult Cardiac Surgical Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG MAN KIN, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.636-T
Record Dates: First submitted 2023-05-26; First posted 2023-06-22 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Chronic; Anesthesia
Keywords: cardiac surgery
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain | interventions — Methadone; Morphine

STUDY DESIGN:
Intervention Model Description: The patients are randomized to receive either methadone 0.2mg/kg (maximum dose of 20mg) or equipotent dose of morphine, added to a syringe containing saline made up to 50ml in total. Randomization will be carried out by an independent investigator, on the day before operation, from pre-prepared envelops each containing the group assignment of either methadone or morphine group. The group assignment will be done by sequence generation with computer models.
Who Masked: Participant, Care Provider
Masking Description: The study syringes containing the drug solution will be of identical appearance and with blind labelling so that the primary care team and the patient will be blinded to the treatments. An independent assessor blinded to the study will be responsible for the data analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Methadone group (Experimental): Upon induction of anaesthesia, intravenous methadone 0.2mg/kg (maximum dose 20mg) in blind labelling will be administered by infusion over 30 minutes. No further morphine will be given throughout the operation, but administration of Intraoperative fentanyl will be left to the discretion of the attending anaesthesiologists
  Interventions: Drug: Methadone
- Morphine group (Active Comparator): Upon induction of anaesthesia, intravenous morphine that is of equipotent dose as 0.2mg/kg methadone or 20mg methadone if maximum dose of interventional drug is reached) in blind labelling will be administered by infusion over 30 minutes. No further morphine will be given throughout the operation, but administration of Intraoperative fentanyl will be left to the discretion of the attending anaesthesiologists
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Methadone — The drug will be prepared by study investigator and then handover to the anaesthesiologist which is blinded to the study. The syringe will be labelled as study drug and given on induction of anaesthesia as intravenous infusion over 30 minutes
  Arms: Methadone group
Drug: Morphine — The drug will be prepared by study investigator and then handover to the anaesthesiologist which is blinded to the study. The syringe will be labelled as study drug and given on induction of anaesthesia as intravenous infusion over 30 minutes
  Arms: Morphine group

SUMMARY:
Despite modern day improvements in pain treatment and availability of different analgesic modalities, suboptimal postoperative pain control remains an issue in cardiac surgical patients. Poorly controlled acute postoperative pain is associated with adverse physiological outcomes that impair the recovery of cardiac surgical patients. It is associated with decreased patient satisfaction, delayed postoperative ambulation, and the development of chronic postsurgical pain (CPSP).

Intravenous opioids such as fentanyl and morphine have been the mainstay of perioperative analgesia for cardiac surgery, either by intermittent boluses by healthcare staff or through a patient-controlled device (PCA). The primary problem with this mechanism of delivery is that significant fluctuations in serum opioid concentrations can occur, resulting in effects which range from inadequate analgesia to overdose and respiratory depression. In contrast to intermittent administration of short-acting opioids such as morphine and fentanyl, a single dose administration of methadone can be considered.

DETAILED DESCRIPTION:
Despite modern day improvements in pain treatment and availability of different analgesic modalities, suboptimal postoperative pain control remains an issue in cardiac surgical patients. Acute postoperative pain is common among cardiac surgical patients, particularly within the first 2 days after surgery, with reported at least moderate intensity. There could be many facets for postoperative pain after adult cardiac surgery. Pain can be caused by surgical incisions and dissections, sternal fracture or incomplete bone healing, multiple drainage cannulas and chest tubes and sternal wound infections. Poorly controlled acute postoperative pain is associated with adverse physiological outcomes that impair the recovery of cardiac surgical patients. It is associated with decreased patient satisfaction, delayed postoperative ambulation, and the development of chronic postsurgical pain (CPSP). The association between sternotomy pain and pulmonary complications has been observed, and the sympathetic activation secondary to pain can induce myocardial ischemia and arrhythmias. Pain control has also been pointed out as one of the major concerns to cardiac surgical patients in intensive care unit. Therefore, optimal acute pain control not only can improve clinical outcomes, but also improves patient satisfaction after cardiac surgery.

Postoperative pain that persists beyond the normal time for tissue healing is increasingly recognized as an important complication after various types of surgery. According to the International Association for Study of Pain, CPSP is defined as the persistence of pain at surgical site or referred area, at least 3 months following the surgical procedure. CPSP is common after cardiac surgery. The reported incidence was 28% to 56% up to 2 years postoperatively. Several mechanisms have been involved in the development of chronic pain after sternotomy. These include dissection, nerve entrapment by sternal wires, sternal retraction, ribs fractures, and intercostal neuralgia as a consequence of nerve damage during dissection of the internal mammary artery during coronary artery bypass graft (CABG). In addition, poorly controlled pain has been a general risk factor for the development of CPSP. All can stimulate the release of pro-inflammatory cytokines which sensitize the afferent nociceptive fibres to cause chronic pain. CPSP has the potential to impact daily functioning and quality of life of patients, as well as increasing the healthcare costs. CARDpain study reported that among those with CPSP, over 50% had significant pain-related interferences with activities of daily living (family and home responsibilities, recreation and employment) at 3, 6 and 12 months following cardiac surgery. Therefore, apart from optimal acute pain control, it is equally important to prevent and manage CPSP, to ensure better satisfaction and quality of lives for our patients.

Intravenous opioids such as fentanyl and morphine have been the mainstay of perioperative analgesia for cardiac surgery, either by intermittent boluses by healthcare staff or through a patient-controlled device (PCA). The primary problem with this mechanism of delivery is that significant fluctuations in serum opioid concentrations can occur, resulting in effects which range from inadequate analgesia to overdose and respiratory depression. These peaks and troughs of analgesia that occur with intermittent opioids administration may explain the suboptimal pain control during the initial postoperative period. In contrast to intermittent administration of short-acting opioids such as morphine and fentanyl, a single dose administration of methadone can be considered. Methadone was conventionally used in cancer and chronic pain management. It can be administered via oral, intravenous, and other parenteral routes. Despite being an often-used alternative to morphine, it remains relatively invisible in perioperative settings. Methadone is a unique opioid that may provide several important potential benefits for surgical patients in the perioperative period. It is a potent mu receptor agonist with a rapid onset and longest half-life (24-36 hours) of the clinically used opioids. According to a pharmacokinetic study, central nervous system effect site methadone concentration rapidly equilibrates with plasma concentrations, evidenced by a short lag time between plasma concentrations and effects (t1/2ke0 4min). This is comparable to the rapid onset and effect compartment equilibration of fentanyl and sulfentanil (5-6min), and in contrast the slow onset time of morphine, where t1/2ke0 has been reported to exceed 4 hours. In addition, as reviewed in an editorial, when methadone is administered at a dose of 20mg or higher, the duration of analgesia approximates the half-life of 24-36 hours. Therefore, a single intravenous dose 20mg administered to an adult at induction of anaesthesia should provide a rapid onset and significant pain relief up to 1-2 days postoperatively, which is the period reported to have the highest pain score after cardiac surgery. Methadone is also a N-methyl-D-aspartate (NMDA) receptor antagonist. It has been reported to possess anti-hyperanalgesic and anti-allodynic properties, that is important in preventing pain sensitization and the development of CPSP, which is of high risk in cardiac surgical patients.

There have been few randomized controlled trials comparing between intravenous methadone and other opioids for perioperative pain control in cardiac surgery requiring sternotomy, and none in the Asian populations. In addition, the effect of methadone on chronic postsurgical pain in cardiac surgical patients has not been widely reported in literature. Therefore, the primary aim of this pilot randomized controlled trial is a feasibility study to evaluate the protocol and the effect of methadone on acute and chronic pain control after open cardiac surgery, compared with conventional approach of opioid-based analgesia using morphine and fentanyl. In addition, the effects of methadone on opioids consumption, opioid-related side effects, patient satisfaction, postoperative extubation times, and length of stay in hospital and ICU will be determined. The investigators hypothesized that intravenous methadone is associated with a reduction in opioids requirement intraoperatively and in the first 24 hours after surgery, and improvement in acute pain score at 12h after extubation. The secondary hypothesis is that patients administered with methadone would experience less CPSP compared with standard treatment group.

The investigators hypothesized that intravenous methadone is feasible and applicable in cardiac anaesthesia, and is associated with opioid-sparing intraoperatively and within 24h after surgery, as well as better acute and chronic pain control when compared to conventional opioid-based approach with morphine and fentanyl in adult cardiac surgical patients. The aims of the study are as follows:

1. To determine the feasibility of using intravenous methadone in adult cardiac surgical patients
2. To evaluate the effect of methadone in acute and chronic pain management in adult cardiac surgical patients requiring sternotomy

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Elective primary isolated coronary artery bypass grafting, aortic valve repair/replacement, mitral valve repair/replacement or combined coronary artery bypass/valve procedure via sternotomy
* Expected extubation within 12 hours of surgery

Exclusion Criteria:

* emergency surgery
* aortic surgery
* redo surgery
* preoperative renal failure requiring renal replacement therapy or creatinine clearance <30ml/min (calculated by Cockcroft-Gault Formula
* liver dysfunction (liver enzymes twice upper limit normal)
* LVEF < 40% at baseline
* mechanical circulatory support in perioperative period
* history of chronic pain or who regularly used pain medications (except paracetamol and non-steroidal anti-inflammatory drugs)
* history of psychiatric illnesses or illicit drug use
* intraoperative use of remifentanil
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients that can be recruited | At recruitment
  defined as the number of patients that fit the recruitment criteria divided by the total number of elective cardiac surgical patients over a period of time
Proportion of patients excluded based on inclusion and exclusion criteria | At recruitment
  Number of patients excluded divided by the total number of elective cardiac surgical patients over a period of time
Cardiac arrhythmia from side effects of methadone | intraoperatively
  New-onset cardiac arrhythmia or prolonged QTc attributed to methadone
Cardiac arrhythmia from side effects of methadone | Within 72 hours postoperatively
  New-onset cardiac arrhythmia or prolonged QTc attributed to methadone

SECONDARY OUTCOMES:
Ventilator time | Within 24 postoperatively in ICU
  The time at which the patient is successfully weaned to spontaneous breathing according to ICU ASV protocol
Total morphine consumption | intraop and postop within 24 hours
  Morphine consumption within 24 hours after operation
Intraoperative fentanyl consumption | intraoperative
  Fentanyl consumption intraoperatively
Pain score at rest | Within 72 hours postop
  Measured using numerical rating scale. It ranges from 0-10. The higher the score, the worse the pain
Pain score on exertion | within 72 hours postop
  Measured using numerical rating scale
Time to first morphine rescue | Postoperatively up to 24 hours
  This is the time the patient feels the need to use morphine from patient-controlled analgesia machine
Nausea and vomiting | Postoperative within 72 hours
  Number of episodes of postoperative nausea and vomiting
Length of hospital stay | upon discharge from hospital (assessed up to day 10)
  Number of hours the patient has to stay in hospital
Length of ICU stay | Upon discharge from ICU (assessed up to day 2)
  Number of hours the patient has to stay in ICU
BPI at 3 months | At 3 months postop
  Measured using Brief Pain Inventory which consists of pain measurement that affects daily living from scale 0-10. The higher the score, the worse the pain
BPI at 6 months | At 6 months postop
  Measured using Brief Pain Inventory which consists of pain measurement that affects daily living from scale 0-10. The higher the score, the worse the pain
NPQ at 3 months | At 3 months postop
  Measured using Neuropathic Pain Questionnaire that has scale 0-100. The higher the score, the worse the pain
NPQ at 6 months | At 6 months postop
  Measured using Neuropathic Pain Questionnaire that has scale 0-100. The higher the score, the worse the pain
PCS at 3 months | At 3 months postop
  Measured using Pain Catastrophizing Scale. It consists of 13 items with each item scaled 0-4. The higher the score, the worse the pain
PCS at 6 months | At 6 months postop
  Measured using Pain Catastrophizing Scale. It consists of 13 items with each item scaled 0-4. The higher the score, the worse the pain

CONTACTS AND LOCATIONS:
Overall Officials: Man Kin WONG, MBChB, Principal Investigator — Chinese Unversity of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Wong HMK, Wong WT, Liu X, Au SSW, Wong RHL. Intravenous methadone for perioperative acute and chronic pain management in Chinese adult cardiac surgical patients: A protocol for pilot randomized controlled trial. PLoS One. 2025 Jun 2;20(6):e0323820. doi: 10.1371/journal.pone.0323820. eCollection 2025. PMID 40455731

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT05913284/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT05913284/ICF_001.pdf